CLINICAL TRIAL: NCT04005638
Title: Biological Bank for the Patients Followed in a Constitutive Reference Center for Autoimmune Cytopenia
Acronym: BIOCAI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry for Health and Solidarity, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/13
Record Dates: First submitted 2019-06-17; First posted 2019-07-02 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Immune Thrombocytopenia; Autoimmune Hemolytic Anemia; Autoimmune Neutropenia
Keywords: Biological collection
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Anemia, Hemolytic, Autoimmune | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 45 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation and urine sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Autoimmune Cytopenia
  Interventions: Biological: blood sample; Biological: urine sample

INTERVENTIONS:
Biological: blood sample — 45 ml whole blood for Peripheral blood mononuclear cell (PBMC) and monocytes isolation
Biological: urine sample — 12 ml

SUMMARY:
The Internal Medicine Department of Haut-Lévêque Hospital (Pr E LAZARO, Pr JL PELLEGRIN, Pr JF VIALLARD) was accredited in 2017 by the Ministry of Health as a Constitutive Reference Center for Autoimmune Cytopenia. The investigators wish to launch new research projects in autoimmune cytopenia and propose a translational and fundamental research based on collaboration between the clinical department, the biological resource center and the CNRS and INSERM research units ("Bedside to the Bench Strategy"). Thus, in the perspective of future research work, it seems imperative to set up a biological bank for the patients followed in our Reference Center.

DETAILED DESCRIPTION:
Our department follows about 350 patients with immune thrombocytopenia (ITP), 50 with autoimmune hemolytic anemia (AHA), and about thirty patients for autoimmune neutropenia and erythroblastopenia. The number of new patients per year is about 50. The investigators are working since several years on different research topics concerning ITP and AHA.

In the field of ITP, the investigators are working on abnormalities of megakaryopoiesis present in a particular subgroup of patients. The investigators seek to identify the molecular mechanisms underlying this platelet-forming disorder. This research is done within the INSERM U1034 unit of the University of Bordeaux.

In AHA, The investigators are working on the role of regulatory CD8+ T lymphocytes and the interest of low doses of Interleukin-2 in their treatment. This part is carried out within the CNRS unit UMR 5164 ImmunoConcept. The biological collection the investigators wish to create will be available for basic research projects and may be available to the pharmaceutical industry as part of the development of new molecules.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 16 years old.
* Patients with autoimmune cytopenia according to the definitions reported in the latest update of the French National Care Protocol (PNDS 2017).
* Affiliated person or beneficiary of a social security scheme.
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Positivity for HIV, Hepatitis C or B virus.
* Pregnant or lactating woman.
* Patient undergoing treatment for autoimmune cytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with autoimmune cytopenia according to the definitions reported in the latest update of the French National Care Protocol (PNDS 2017).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-02-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with autoimmune cytopenia at diagnosis, or followed but not treated with a biological library (serum, plasma, DNA) | At baseline (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François VIALLARD, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service de médecine interne, Pessac, France

IPD SHARING:
Plan to Share IPD: No